CLINICAL TRIAL: NCT06417372
Title: Prospective Study of the Effect of Intraoperative Fluorescent Staining Combined With Microscopy on the Prognosis of Patients With Gliomas
Brief Title: Intraoperative Fluorescent Staining Combined With Microsurgery for Gliomas
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhang Nu, Discipline Leader of Neurosurgery department, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2023]670-FM
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Glioma
Keywords: glioma
MeSH Terms: conditions — Glioma | interventions — Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: 1. any gender, age 18-60 years old;
  2. patients with a confirmed diagnosis of glioma (primary tumor or metastatic tumor) by imaging or biopsy;
  3. patients who can tolerate the surgery by preoperative evaluation; the expected volume of tumor specimen to be resected intraoperatively is more than 1cm3;
  4. subjects who voluntarily enroll in the study, sign the informed consent form, and have a good adherence to the study and cooperate with the follow-up visits;
  5. patients with expected survival of not less than 12 months as judged by clinician; and 6. patients who are not in the clinical trial. The expected survival period, as judged by the clinician, is not less than 12 months.
  Interventions: Diagnostic Test: intraoperative fluorescent staining combined with microscopy

INTERVENTIONS:
Diagnostic Test: intraoperative fluorescent staining combined with microscopy — Through the modified formulation of sodium fluorescein and methylene blue, the surface of the suspected cut edge of the patient's glioma was stained intraoperatively, and the surgical microscope image acquisition and processing system was used to determine whether the cut edge of the surgically resected tissue was positive or not.

SUMMARY:
Through the modified formulation of sodium fluorescein and methylene blue, the surface of the suspected cut edge of the patient's glioma was stained intraoperatively, and the surgical microscope image acquisition and processing system was used to determine whether the cut edge of the surgically resected tissue was positive or not. And combined with the existing multimodal surgical techniques (imaging, electrophysiology, neuronavigation and other equipment), the glioma is precisely resected.

ELIGIBILITY:
Inclusion Criteria:

1. any gender, age 5-90 years old;
2. patients with a confirmed diagnosis of glioma (primary tumor or metastatic tumor) by imaging or biopsy;
3. patients who can tolerate the surgery by preoperative evaluation; the expected volume of tumor specimen to be resected intraoperatively is more than 1cm3;
4. subjects who voluntarily enroll in the study, sign the informed consent form, and have a good adherence to the study and cooperate with the follow-up visits;
5. patients with expected survival of not less than 12 months as judged by clinician; and 6. patients who are not in the clinical trial. The expected survival period, as judged by the clinician, is not less than 12 months.

Exclusion Criteria:

1. Serious or unstable diseases of the heart, lungs, kidneys and hematopoietic system that cannot tolerate surgery
2. Pregnant or lactating women
3. Other factors that, in the judgment of the investigator, could lead to termination of the study, such as other serious medical conditions or serious laboratory abnormalities or other family or social factors that would affect the safety of the subject or the collection of test data and samples.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed glioma patients who will undergo surgical treatment in the First Affiliated Hospital of Sun Yet-Sen Universtiy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | From date of randomization until the date of first documented progression, assessed up to 12 months
  progression-free survival (PFS): From date of randomization until the date of first documented progression
overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 18 months
  overall survival (OS): From date of randomization until the date of death from any cause